CLINICAL TRIAL: NCT02136979
Title: Effect of Propofol and Sevoflurane on Serum CD39 and CD73 Level After Open Heart Surgery With Cardiopulmonary Bypass
Brief Title: Effect of Anesthetics on CD39 and CD73 After Open-heart Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Hyop Kim, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: KUH1160064
Record Dates: First submitted 2014-05-07; First posted 2014-05-13 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Valvular Heart Disease; Aortic Disease
MeSH Terms: conditions — Heart Valve Diseases; Aortic Diseases | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol group (Active Comparator): patients with propofol-based anesthesia
  Interventions: Drug: Propofol
- Sevoflurane group (Active Comparator): patients with sevoflurane-based anesthesia
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — group of patients with propofol-based anesthesia
  Other Names: Propofol group
  Arms: Propofol group
Drug: Sevoflurane — group of patients with sevoflurane-based anesthesia
  Other Names: Sevoflurane group
  Arms: Sevoflurane group

SUMMARY:
CD39 and CD73 was known protein expressed on surface of Th1 and Th17 cell and modulate immune related reaction. Cardiopulmonary bypass (CPB) can induce inflammatory reaction during cardiac surgery, and induce immunosuppression. Propofol and volatile anesthetics were related to immune reaction. However, the effect of propofol and sevoflurane on the change of CD39 and CD73 after CPB was not evaluated in previous studies.

The authors hypothesized that the expression of CD39 and CD73 would differ between propofol- and volatile anaesthetic-based anaesthesia in patients undergoing CPB. Therefore, the present study determined the effect of propofol and sevoflurane on CD39 and CD73 during and after CPB.

DETAILED DESCRIPTION:
After obtaining permission of the Institutional Review Board of Konkuk University Medical Center, Seoul, South Korea , patients scheduled to undergo elective cardiac surgery under cardiopulmonary bypass (CPB) after signed written informed consent agreements and prospectively participate in the present study.

All patients got a cardiac surgery under moderate hypothermic cardiopulmonary bypass (CPB) by one cardiac surgeon. Also, 6ml of blood and sample was obtained for total 5 times in consecutive order.

1. Before operation (pre-CPB1)
2. 15 minute after successful CPB weaning (post-CPB1)
3. 3 hrs after CPB weaning (post-CPB2)
4. 24 hrs after CPB weaning (post-CPB3)
5. 48 hrs after CPB weaning (post-CPB4)

The following intraoperative exclusion criteria are applied:

1. Emergency operation that could not obtain pre-CPB1 sample
2. Patients who have infectious factor before operation
3. Patients who have immunosuppressive agent for underlying disease before operation
4. Patients who have history of cancer previously
5. Patients who are younger than 19 years old

Using blood sample, authors examined as follows

1. Flow cytometry for Th 17 and Th 1 cell.
2. Immunocytochemistry for CD39, CD73.
3. Assay for IL 1,6,10,17,IFN-γ, and TNF-α
4. patient vital sign during operation
5. other laboratory tests

Statistical analyses are conducted using SPSS 20.0 (SPSS Inc., Chicago, IL, USA). CD39 and CD73 are analysed used a Repeated Measures Analysis of Variance and their pairwise multiple comparisons are performed via the tukey method. The comparisons of the other continuous variables are performed by paired t or Wilcoxon Signed Rank tests. Data are expressed as mean ± SD (95% confidence interval. CI) or median (25%-75%), and number of the patients. A p value less than 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. patients scheduled to undergo elective cardiac surgery
2. signed written informed consent agreements

Exclusion Criteria:

1. Emergency operation that could not obtain pre-CPB1 sample
2. Patients who have infectious factor before operation
3. Patients who have immunosuppressive agent for underlying disease before operation
4. Patients who have history of cancer previously
5. Patients who are younger than 19 years old

Ages: 19 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
The level of CD39 and CD73 between propofol and sevoflurane group after CPB | from preoperative status up to 48 hrs after CPB weaning status
  The difference of CD39 and CD73 level between propofol and sevoflurane group

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D, Ph.D, Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea